CLINICAL TRIAL: NCT05215340
Title: A Randomized, Open-label, Phase 3 Trial of Dato-DXd Plus Pembrolizumab vs Pembrolizumab Alone in Treatment-naïve Subjects With Advanced or Metastatic PD-L1 High (TPS ≥50%) Non-small Cell Lung Cancer Without Actionable Genomic Alterations (TROPION-Lung08)
Brief Title: Study of Dato-DXd Plus Pembrolizumab vs Pembrolizumab Alone in the First-line Treatment of Subjects With Advanced or Metastatic NSCLC Without Actionable Genomic Alterations
Acronym: TROPION-Lung08
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Daiichi Sankyo (Industry)
Collaborators: AstraZeneca (Industry); Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DS1062-A-U304; 2021-002555-10 (EudraCT Number); KEYNOTE-C73 (Other: Merck); MK3475-C73 (Other: Merck); 2023-507933-12-00 (EU CTIS Number)
Record Dates: First submitted 2022-01-18; First posted 2022-01-31 (Actual); Last update posted 2026-01-07 (Actual); Status verified 2026-01

CONDITIONS: Metastatic Non Small Cell Lung Cancer
Keywords: Metastatic Non Small Cell Lung Cancer; Advanced Non Small Cell Lung Cancer; Datopotamab Deruxtecan (Dato-DXd); Pembrolizumab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Datopotamab Deruxtecan (Dato-DXd) (Experimental): Participants will be randomized to receive 200 mg pembrolizumab followed by 6.0mg/kg Dato-DXd.
  Interventions: Drug: Datopotamab Deruxtecan; Drug: Pembrolizumab
- Pembrolizumb (Active Comparator): Participants will be randomized to receive 200 mg pembrolizumab.
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: Datopotamab Deruxtecan — Dato-DXd will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Other Names: Dato-DXd
  Arms: Pembrolizumab + Datopotamab Deruxtecan (Dato-DXd)
Drug: Pembrolizumab — Pembrolizumab will be administered as an intravenous (IV) infusion every 3 weeks on Day 1 of each 21-day cycle.
  Other Names: KEYTRUDA®

SUMMARY:
This study is designed to assess the efficacy and safety of datopotamab deruxtecan (Dato-DXd) in combination with pembrolizumab versus pembrolizumab alone in participants with advanced or metastatic non-small cell lung cancer (NSCLC) of non-squamous histology.

DETAILED DESCRIPTION:
The primary objective of the study is to compare the efficacy of Dato-DXd and pembrolizumab with pembrolizumab alone in terms of either Progression Free Survival (PFS) by BICR or Overall Survival (OS) for participants with advanced or metastatic NSCLC with non-squamous histology without actionable genomic alterations whose tumor has high programmed death-ligand 1 (PD-L1) expression (tumor proportion score; TPS ≥50%) and who have not previously received systemic therapy for advanced or metastatic NSCLC.

Eligible participants will be randomized in a 1:1 ratio to the control arm (pembrolizumab alone) or the experimental arm (Dato-DXd and pembrolizumab). The study will be divided into 4 periods: Tissue Screening Period, Screening Period, Treatment Period, and Follow-up Period.

ELIGIBILITY:
Inclusion Criteria:

Participants eligible for inclusion in the study must meet all inclusion criteria within 28 days of randomization into the study.

* Sign and date the Tissue Screening and Main Informed Consent Forms, prior to the start of any study-specific qualification procedures.
* Adults ≥18 years or the minimum legal adult age (whichever is greater) at the time of informed consent.
* Histologically documented non-squamous NSCLC that meets all of the following criteria (Note: Subjects with squamous histology were eligible prior to Protocol Version 5.0. After Protocol Version 5.0, subjects with squamous histology are not eligible. Subjects with mixed histology, including those with a squamous component, remain eligible the study even after Protocol Version 5.0):

  1. Stage IIIB or IIIC disease and not candidates for surgical resection or definitive chemoradiation, or Stage IV NSCLC disease at the time of randomization (based on the American Joint Committee on Cancer, Eighth Edition). Participants with early-stage NSCLC who have relapsed should be restaged during screening to ensure their eligibility for the study.
  2. Documented negative test results for epidermal growth factor receptor (EGFR), lymphoma kinase (ALK), and proto-oncogene1 (ROS1) actionable genomic alterations (AGAs) based on analysis of tumor tissue. If test results for EGFR, ALK, and ROS1 are not available, subjects are required to undergo testing performed locally for these genomic alterations.
  3. No known AGAs in neurotrophic tyrosine receptor kinase (NTRK), proto-oncogene B-raf (BRAF), rearranged during transfection (RET), mesenchymal-epithelial transition factor (MET), or other actionable driver kinases with locally approved therapies. (Testing for genomic alterations besides EGFR, ALK, and ROS1 is not required prior to randomization). Subjects whose tumors harbor KRAS mutations are eligible for the study.
* Has provided a formalin-fixed tumor tissue sample for the measurement of trophoblast cell surface protein 2 (TROP2) protein expression and for the assessment of other exploratory biomarkers.
* Tumor has high programmed death receptor-1 (PD-L1) expression (TPS ≥50%) as determined by PD-L1 immunohistochemistry (IHC) 22C3 pharmDx assay by central testing (minimum of 6 slides).
* Has an adequate treatment washout period before Cycle 1 Day 1.
* Measurable disease based on local imaging assessment using RECIST Version 1.1.
* Has left ventricular ejection fraction (LVEF) ≥50% by either an echocardiogram (ECHO) or multigated acquisition scan (MUGA) within 28 days before randomization.
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) of 0 or 1 at screening.
* Has a life expectancy of at least 3 months.
* Adequate bone marrow function within 7 days before randomization.

Exclusion Criteria:

* Has received prior systemic treatment for advanced or metastatic NSCLC.
* Has received prior treatment for NSCLC with any of the following, including in the adjuvant/neoadjuvant setting:

  1. Any agent, including an antibody-drug conjugate, containing a chemotherapeutic agent targeting topoisomerase I.
  2. TROP2-targeted therapy.
  3. Any anti-programmed death receptor-1 (PD-1), anti-PD-L1, or anti-PD-ligand 2 (L2) agent or with an agent directed to another stimulatory or co-inhibitory T-cell receptor (eg, CTLA-4, OX40, CD137).
  4. Any other immune checkpoint inhibitors. Participants who received adjuvant or neoadjuvant therapy OTHER than those listed above, are eligible if the adjuvant/neoadjuvant therapy was completed at least 6 months prior to the diagnosis of advanced/metastatic disease.
* Has spinal cord compression or active and untreated central nervous system (CNS) metastases and/or carcinomatous meningitis. Participants with previously treated brain metastases and who are asymptomatic may participate provided they are radiologically stable.
* Has received prior radiotherapy < 4 weeks of start of study intervention or more than 30 Gy (unit of ionizing radiation dose in the International System of Units) to the lung within 6 months of Cycle 1 Day 1.
* History of another primary malignancy (beyond NSCLC) except for:

  1. Malignancy treated with curative intent and with no known active disease ≥3 years before the first dose of study treatment and of low potential risk for recurrence.
  2. Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease.
  3. Adequately treated carcinoma in situ without evidence of disease.
  4. Participants with a history of prostate cancer (tumor/node/metastasis stage) of Stage ≤T2cN0M0 without biochemical recurrence or progression and who in the opinion of the Investigator are not deemed to require active intervention.
* Has a history of (non-infectious) interstitial lung disease (ILD)/pneumonitis including radiation pneumonitis that required steroids, has current ILD/pneumonitis, or where suspected ILD/pneumonitis cannot be ruled out by imaging at screening.
* Clinically severe pulmonary compromise, as judged by the investigator, resulting from intercurrent pulmonary illnesses including, but not limited to, any underlying pulmonary disorder, or any autoimmune, connective tissue or inflammatory disorders with pulmonary involvement or prior complete pneumonectomy.
* Uncontrolled or significant cardiovascular disease, including:

  1. Mean QT interval corrected for heart rate using Fridericia's formula (QTcF) interval >470 ms regardless of sex (based on the average of the 12-lead electrocardiogram determination at screening).
  2. Myocardial infarction within 6 months prior to randomization.
  3. Uncontrolled angina pectoris within 6 months prior to randomization.
  4. LVEF <50% by ECHO or MUGA scan within 28 days before randomization.
  5. New York Heart Association Class 2 to 4 congestive heart failure (CHF) at screening.
  6. Uncontrolled hypertension (resting systolic blood pressure >180 mmHg or diastolic blood pressure >110 mmHg) within 28 days before randomization.

Participants with a history of Class 2 to 4 CHF prior to screening, must have returned to Class 1 CHF and have LVEF ≥50% (by either an ECHO or MUGA scan within 28 days before randomization) in order to be eligible.

* Clinically significant corneal disease.
* Has received a live vaccine or live-attenuated vaccine (messenger ribonucleic acid and replication-incompetent adenoviral vaccines are not considered attenuated live vaccines) within 30 days prior to the first dose of study drug. For any participant receiving an approved severe acute respiratory syndrome coronavirus 2 (SARS-CoV2) vaccine, please follow the vaccine label and/or local guidance.
* Active, known, or suspected autoimmune disease (has an active autoimmune disease that has required systemic treatment in the past 2 years).
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosage >10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy ≤7 days prior to the first dose of study drug.
* Has known human immunodeficiency virus (HIV) infection that is not well controlled.
* Has an active hepatitis or uncontrolled hepatitis B or active hepatitis C infection.
* Has an uncontrolled infection requiring IV antibiotics, antivirals, or antifungals.
* Had an allogeneic tissue/solid organ transplant.
* Has a history of severe hypersensitivity reactions to either the drug or inactive ingredients (including but not limited to polysorbate 80) of Dato-DXd or pembrolizumab.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 740 (Estimated)
Dates: Start 2022-03-04 (Actual); Primary Completion 2028-02-29 (Estimated); Study Completion 2028-04-30 (Estimated)

PRIMARY OUTCOMES:
Progression-free Survival Based on Blinded Independent Central Review in Participants With Non-Squamous Histology Who Were Administered Dato-DXd in Combination With Pembrolizumab Compared With Pembrolizumab | From randomization until disease progression or death (whichever occurs first), up to approximately 44 months
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by blinded independent central review (BICR) per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
Overall Survival (OS) in Participants With Non-Squamous Histology Who Were Administered Dato-DXd in Combination With Pembrolizumab Compared With Pembrolizumab | From randomization until date of death due to any cause, up to approximately 71 months
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.

SECONDARY OUTCOMES:
OS in All Randomized Participants, Including Participants With Squamous and Non-Squamous Histology | From randomization until date of death due to any cause, up to approximately 71 months
  Overall Survival (OS) is defined as the time from randomization to death due to any cause.
PFS Based on BICR in All Randomized Participants, Including Participants With Squamous and Non-Squamous Histology | From randomization until disease progression or death (whichever occurs first), up to approximately 44 months
  PFS is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by BICR per Response Evaluation Criteria in Solid Tumors (RECIST), Version 1.1.
Progression-free Survival by Investigator in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization until disease progression or death (whichever occurs first), up to approximately 44 months
  Progression-free Survival (PFS) is defined as the time from randomization to the first documented radiographic disease progression or death due to any cause, whichever occurs first, assessed by the Investigator per RECIST Version 1.1.
Progression-free Survival 2 in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization until disease progression on the next line of therapy or death (whichever occurs first), up to approximately 71 months
  Progression-free Survival 2 (PFS2) is defined as the time from date of randomization to the first documented disease progression on next-line therapy or death due to any cause, whichever occurs first.
ORR by BICR and Investigator in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization to first confirmed response, up to approximately 44 months
  Objective Response Rate (ORR) is defined as the proportion of participants who achieved a best overall response (BOR) of confirmed complete response (CR) or confirmed partial response (PR), assessed by BICR and by the Investigator per RECIST Version 1.1.
Duration of Response by BICR and Investigator in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From date of first objective response (CR or PR) to date of first radiographic disease progression or death due to any cause (whichever occurs first), up to approximately 44 months
  Duration of Response (DoR) is defined as the time from the date of the first documentation of objective response (confirmed CR or confirmed PR) to the date of the first radiographic disease progression or death due to any cause, whichever occurs first, assessed by BICR and by the Investigator per RECIST Version 1.1.
Time to Response by BICR and Investigator in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization to date of first objective response (CR or PR), up to approximately 44 months
  Time to Response (TTR) is defined as the time from randomization to the date of the first documentation of objective response (confirmed CR or confirmed PR) in responding participants, assessed by BICR and by the Investigator per RECIST Version 1.1.
Disease Control Rate by BICR and Investigator in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization until disease progression or death (whichever occurs first), up to approximately 44 months
  Disease Control Rate (DCR) is defined as the proportion of participants who achieved a BOR of confirmed CR, confirmed PR, or stable disease (SD), assessed by BICR and by the Investigator per RECIST Version 1.1.
Time to Deterioration in Participants with Non-Squamous Histology, and Separately for All Randomized Participants | From randomization until disease progression or death (whichever occurs first), up to 71 months
  Time to Deterioration (TTD) is defined as the time from randomization to first onset of a ≥10-point increase in cough, chest pain, or dyspnea, confirmed by a second adjacent ≥10-point increase from randomization in the same symptom, or confirmed by death within 21 days of a ≥10-point increase from randomization, assessed the European Organization for Research and Treatment of Cancer Lung cancer module (EORTC-QLQ-LC13).
Number of Participants With Treatment-emergent Adverse Events (TEAE) with Non-Squamous Histology, and Separately for All Randomized Participants | Up to 71 months
  A TEAE is defined as an AE with a start or worsening date on or after the start date of study treatment until 37 days after the end date of study treatment.
Proportion of Participants Who Are Anti-Drug Antibody (ADA)-Positive (Baseline and Post-Baseline) and Proportion of Participants Who Have Treatment-emergent ADA for Participants with Non-Squamous Histology, and Separately for All Randomized Participants | Baseline and up to 71 months
  The immunogenicity of Dato-DXd in combination with pembrolizumab will be assessed.

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Leader, Study Director — Daiichi Sankyo
Locations (243):
- United States (36):
  - Ironwood Cancer and Research Center, Chandler, Arizona
  - UCLA HemOnc - Clinical Research Unit, Los Angeles, California
  - Compassionate Cancer Care Medical Group, Riverside, California
  - UCSF Helen Diller Family Comprehensive Cancer Center, San Francisco, California
  - Ridley-Tree Cancer Center, Santa Barbara, California
  - PIH Health Whittier Hospital, Whittier, California
  - The Oncology Institute of Hope and Innovation, Whittier, California
  - Uch-Mhs D/B/A Memorial Health System, Colorado Springs, Colorado
  - Johns Hopkins University, Baltimore, Maryland
  - American Oncology Partners of Maryland, Bethesda, Maryland
  - Dana-Farber Cancer Institute, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - DFCI - Steward St. Elizabeth's Medical Center, Boston, Massachusetts
  - Dana Farber Cancer Institute - Foxborough, Foxborough, Massachusetts
  - Dana Farber Cancer Institute - Milford Medical Center, Milford, Massachusetts
  - DFCI - South Shore Hospital, South Weymouth, Massachusetts
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Astera Cancer Care, East Brunswick, New Jersey
  - Regional Cancer Care Associates LLC, Freehold, New Jersey
  - Cooperman Barnabas Medical Center, New Brunswick, New Jersey
  - The Valley Hospital, Paramus, New Jersey
  - Montefiore Medical Center, The Bronx, New York
  - Arizona Oncology NAHOA, Irving, Texas
  - Cancer Care Center of Brevard, Irving, Texas
  - Illinois Cancer Specialists, Irving, Texas
  - Maryland Oncology Hematology, Irving, Texas
  - Southern Cancer Center, Irving, Texas
  - Texas Oncology - Northeast Texas, Irving, Texas
  - Texas Oncology Gulf Coast, Irving, Texas
  - Texas Oncology McAllen, Irving, Texas
  - Woodlands Medical, Irving, Texas
  - University of Texas Health Science Center San Antonio, San Antonio, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Providence Regional Cancer System, Lacey, Washington
  - VA Puget Sound Health Care System - VAPSHCS, Seattle, Washington
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Argentina (9):
  - Centro de Investigaciones Medicas y Desarrollo LC S.R.L. (LC Investigacion), Buenos Aires
  - Fundacion CENIT para la investigación en Neurociencias, Ciudad Autonoma de Buenos Aire
  - Hospital Privado de la Comunidad, Mar del Plata
  - Centro de Investigación Pergamino S. A., Pergamino
  - Instituto de Oncología de Rosario, Rosario
  - Sanatorio Parque, Rosario
  - Sanatorio Británico de Rosario, Rosario
  - CER SAN JUAN - Centro Polivalente de Asistencia e Investigación Clínica, San Juan
  - Clinica Viedma SA, Viedma
- Australia (4):
  - Austin Hospital, Heidelberg, Victoria
  - Peninsula and South Eastern Haematology and Oncology Group, Mount Waverley, Victoria
  - Chris Obrien Lifehouse, Camperdown
  - The Queen Elizabeth Hospital, Woodville South
- Austria (2):
  - Klinikum Klagenfurt am Wörthersee Abteilung für Lungenkrankheiten, Klagenfurt
  - Karl-Landsteiner Institute for Lung Research and Pulmonary Oncology c/o Klinik Floridsdorf, Vienna
- Belgium (4):
  - Onze-Lieve-Vrouwziekenhuis Olvz - Campus Aalst, Aalst
  - Grand Hopital de Charleroi - Hopital Saint Joseph, Charleroi
  - Az Maria Middelares - Campus Maria Middelares, Ghent
  - AZ Nikolaas, Sint-Niklaas
- Brazil (10):
  - Instituto de Pesquisas em Saúde - IPS, Caxias do Sul
  - Hospital Erasto Gaertner, Curitiba
  - Oncosite - Centro de Pesquisa Clinica Oncologia, Ijuí
  - Clínica de Neoplasias Litoral, Itajaí
  - UPCO - Unidade de Pesquisas Clínicas em Oncologia - Clinica Lacks, Pelotas
  - Santa Casa de Misericordia de Porto Alegre, Porto Alegre
  - Instituto Nacional de Câncer - INCA, Rio de Janeiro
  - Centro de Estudos e Pesquisa de Hematologia e Oncologia - CEPHO, Santo André
  - Instituto de Ensino e Pesquisas Sao Lucas, São Paulo
  - Instituto do Cancer Brasil - Unidade Taubate, Taubaté
- Canada (2):
  - Santa Cabrini Hospital, Montreal
  - McGill University Health Centre, Montreal
- Chile (5):
  - Centro de Estudios Clínicos SAGA, Santiago, Santiago Metropolitan
  - Oncovida, Santiago
  - Fundación Arturo Pérez López, Santiago
  - Orlandi Oncología, Santiago
  - Centro de Investigaciones Clinicas Vina Del Mar, Viña del Mar
- China (32):
  - Guangxi Medical University Affiliated Tumor Hospital, Nanning, Guangxi
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Jilin Cancer Hospital, Changchun, Jilin
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Peking University Peoples Hospital, Beijing
  - Peking University Cancer Hospital, Beijing
  - Cangzhou People's Hospital, Cangzhou
  - Hunan Cancer Hospital, Changsha
  - Army Medical Center of PLA, Chongqing
  - Affiliated Cancer Hospital and Institute of Guangzhou Medical University, Guangzhou
  - Haikou People's Hospital, Haikou
  - The First Affiliated Hospital of College of Medicine Zhejiang University, Hanghzou
  - Zhejiang Cancer Hospital, Hangzhou
  - Harbin Medical University Cancer Hospital, Harbin
  - Inner Mongolia Medical University- the Affiliated Hospital, Hohhot
  - Jiamusi Tumor and Tuberculosis Hospital, Jiamusi
  - Yunnan Cancer Hospital, Kunming
  - Linyi Cancer Hospital, Linyi
  - The First Affiliated Hospital of Nanchang University, Nanchang
  - Jiangsu Province Hospital, Nanjing
  - The Second People's Hospital of Neijiang, Neijiang
  - Shanghai Pulmonary Hospital, Shanghai
  - Fudan University Shanghai Cancer Center, Shanghai Shi
  - The First Hospital of China Medical University, Shenyang
  - Liaoning Cancer Hospital& Institute, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - Xinjiang Tumor Hospital, Ürümqi
  - Union Hospital Affiliated With Tongji Medical College Huazhong University of Science and Technology, Wuhan
  - Hubei Cancer Hospital, Wuhan
  - The First Affiliate Hospitalof Xi'An Jiaotong University, Xi'an
  - The First Affiliated Hospital Xiamen University, Xiamen
  - Xiangyang Central Hospital- 5 Lumen Avenue, Xiangyang
- France (13):
  - Sainte-Catherine Institut du Cancer Avignon-Provence (ICAP), Avignon
  - Bordeaux University Hospital - Hopital Saint Andre, Bordeaux
  - Institut Bergonie, Bordeaux
  - Centre Hospitalier Universitaire de Lille, Lille
  - Centre Leon Berard, Lyon
  - APHM - Hopital Nord, Marseille
  - Institut Paoli-Calmettes, Marseille
  - Centre Hospitalier Universitaire de Montpellier, Montpellier
  - CHU de Nantes, Nantes
  - Hopital prive du Confluent, Nantes
  - AP-HP - Hopital Tenon, Paris
  - CHU de Poitier Pole Regional de Cancerologie, Poitiers
  - Hopital FOCH, Suresnes
- Germany (4):
  - Evangelische Lungenklinik Berlin, Berlin
  - Klinikum Esslingen GmbH, Esslingen am Neckar
  - LungenClinic Grosshansdorf, Großhansdorf
  - Klinikum der Universitaet Muenchen, München
- Greece (7):
  - Metropolitan Hospital, Neo Faliro, Athens
  - Sotiria General Hosptial of Chest Diseases, Athens
  - University Hospital of Ioannina Uhi, Ioannina
  - Metropolitan Hospital, Neo Faliro
  - Metropolitan Hospital, Piraeus
  - Bioclinic Thessaloniki, Thessaloniki
  - St. Luke's Hospital, Thessaloniki
- Hong Kong (3):
  - Prince of Wales Hospital / The Chinese University of Hong Kong 99999, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Pok Fu Lam
- Hungary (5):
  - Semmelweis University Department of Pulmonology, Budapest
  - Veszprem Megyei Tudogyogyintezet Farkasgyepu, Farkasgyepű
  - Bkmk Hospital, KecskemĂŠt
  - Fejer Megyei Szent Gyorgy Egyetemi Oktato Korhaz, Székesfehérvár
  - Pulmonology Hospital Torokbalint, Törökbálint
- Italy (10):
  - IRCCS Istituto Oncologico Giovanni Paolo II, Bari
  - UOC Oncologia, Chieti
  - Ospedale San Luca, Lucca
  - IRCCS Ospedale San Raffaele, Milan
  - Irccs Istituto Europeo Di Oncologia, Milan
  - Azienda Ospedaliera dei Colli, Naples
  - A.O. Perugia Santa Maria della Misericordia, Perugia
  - Policlinico Tor Vergata, Rome
  - Ifo Regina Elena, Rome
  - Asst Sette Laghi Ospedale di Circolo e Fondazione Macchi, Varese
- Japan (27):
  - Aomori Prefectural Central Hospital, Aomori, Aomori
  - National Cancer Center Hospital East, Kashiwa-shi, Chiba
  - NHO Shikoku Cancer Center, Matsuyama, Ehime
  - National Hospital Organization Kyushu Cancer Center, Fukuoka, Fukuoka
  - Kyushu University Hospital, Fukuoka, Fukuoka
  - Kurume University Hospital, Kurume-shi, Fukuoka
  - Kanazawa University Hospital, Kanazawa, Ishikawa-ken
  - Kanagawa Cancer Center, Yokohama, Kanagawa
  - Saiseikai Kumamoto Hospital, Kumamoto, Kumamoto
  - Matsusaka Municipal Hospital, Matsusaka-shi, Mie-ken
  - Sendai Kousei Hospital, Sendai, Miyagi
  - Niigata Cancer Center Hospital, Niigata, Niigata
  - Kansai Medical University Hospital, Hirakata-shi, Osaka
  - Osaka International Cancer Institute, Osaka, Osaka
  - NHO Kinki-Chuo Chest Medical Center, Sakai-shi, Osaka
  - Saitama Cancer Center, Ina-machi, Saitama
  - Dokkyo Medical University Hospital, Shimotsuga-gun, Tochigi
  - Juntendo University Hospital, Bunkyo-ku, Tokyo
  - Tokyo Metropolitan Cancer and Infectious Diseases Center Komagome Hospital, Bunkyō-Ku, Tokyo
  - The Cancer Institute Hospital of JFCR, Kōtoku, Toyko
  - Toho University Omori Medical Center, Ōta-ku, Toyko
  - NHO Iwakuni Clinical Center, Iwakuni-shi, Yamaguchi
  - Yamaguchi-Ube Medical Center, Ube-shi, Yamaguchi
  - Yamanashi Prefectural Central Hospital, Kofu
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Osaka Toneyama Medical Center, Osaka
  - Teine Keijinkai Hospital, Sapporo
- Mexico (5):
  - Cryptex Investigacion Clinica Sa de Cv, Cuauhtémoc
  - Hospital Civil de Guadalajara Fray Antonio Alcalde, Guadalajara
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey
  - Centro de Investigacion Clinica de Oaxaca (CICLO), Oaxaca City
  - Oncologico Potosino, San Luis Potosí City
- Netherlands (4):
  - Rijnstate Ziekenhuis, Arnhem, Gelderland
  - Jeroen Bosch Ziekenhuis J BZ Hieronymus Bosch Hospital, 's-Hertogenbosch
  - Amsterdam Umc, Location Vumc, Amsterdam
  - Leiden University Medical Center, Leiden
- Poland (5):
  - Instytut Centrum Zdrowia Matki Polki, Lodz, Iodzkie
  - Szpitale Pomorskie Sp. z o.o., Gdynia, Pomeranian Voivodeship
  - Dom Lekarski SA, Szczecin, West Pomeranian Voivodeship
  - II Klinika Chorob Pluc I Gruzlicy, Bialystok
  - MS Pneumed Janusz Milanowski, Katarzyna Szmygin-Milanowska Sp. Jawna, Lublin
- Portugal (5):
  - Centro Clinico Champalimau, Lisbon
  - Centro Hospitalar e Universitário do Porto, Porto
  - Hospital CUF Porto, Porto
  - Instituto Portuguas de Oncologia do Porto Francisco Gentil, Porto
  - Centro Hospitalar Universitário de São João, Porto
- Romania (5):
  - Onco Clinic Consult SA, Craiova
  - Centrul de Oncologie Sf Nectarie S.R.L., Craiova
  - Sc Sigmedical Services Srl, Suceava
  - Oncocenter-Oncologie Clinica SRL, Timișoara
  - SC Oncomed SRL, Timișoara
- South Korea (8):
  - Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do
  - Gyeongsang National University Hospital, Jinju, Gyeongsangnam-do
  - Chungbuk National University Hospital, Cheongju-si, North Chungcheong
  - Kyungpook National University Chilgok Hospital, Daegu
  - National Cancer Center, Goyang-si
  - Samsung Medical Center, Seoul
  - The Catholic Univ. of Korea, Seoul St. Mary'S Hospital, Seoul
  - Asan Medical Center, Songpa-gu
- Spain (12):
  - Hospital Clinic i Provincial de Barcelona, Barcelona
  - Hospital Universitari Vall D'Hebron, Barcelona
  - Hospital Universitario Arnau de Vilanova - Lleida, Lleida
  - Hospital General Universitario Gregorio Marañon, Madrid
  - Hospital Clinico San Carlos, Madrid
  - Hospital Universitario Fundacion Jimenez Diaz, Madrid
  - Hospital Regional Universitario Malaga, Málaga
  - CHUO, Ourense
  - Hospital Universitario Virgen Macarena, Seville
  - Hospital Universitario de Valme, Seville
  - Hospital Universitari i Politècnic La Fe, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Switzerland (4):
  - Kantonsspital Baden, Baden
  - University Hospital Basel, Basel
  - Kantonsspital Baselland, Liestal
  - Kantonsspital St. Gallen, Sankt Gallen
- Taiwan (9):
  - E-Da Hospital, Kaohsiung City
  - Chang Gung Memorial Hospital Cgmh - Kaohsiung Branch, Kaohsiung City
  - Chung Shan Medical University Hospital, Taichung
  - Taichung Veterans General Hospital, Taichung
  - National Cheng Kung University Hospital Nckuh, Tainan
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
  - Koo Foundation Sun Yat-Sen Cancer Center, Taipei
  - Chang Gung Memorial Hospital LinKou, Taoyuan District
- Thailand (4):
  - Srinagarind Hospital, Muaeng, Changwat Khon Kaen
  - Prince of Songkla University PSU - Faculty of Medicine, Hat Yai, Changwat Songkhla
  - Faculty of Medicine Chulalongkorn University, Bangkok
  - Siriraj Hospital, Bangkok
- Turkey (Türkiye) (6):
  - Adana Acibadem Hospital, Adana
  - Akdeniz University Hospital, Antalya
  - Ege University, Bornova-İzmir
  - Memorial Ankara Hospital Ankara, Çankaya
  - Goztepe Prof. Dr. Suleyman Yalcin City Hospital, Istanbul
  - Medical Park Seyhan Hospital, Seyhan /Adana
- United Kingdom (3):
  - Birmingham Heartlands Hospital, Birmingham
  - Beatson West of Scotland Cancer Centre, Glasgow
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data (IPD) and applicable supporting clinical trial documents may be available upon request at https://vivli.org/. In cases where clinical trial data and supporting documents are provided pursuant to our company policies and procedures, Daiichi Sankyo will continue to protect the privacy of our clinical trial participants. Details on data sharing criteria and the procedure for requesting access can be found at this web address: https://vivli.org/ourmember/daiichi-sankyo/
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Studies for which the medicine and indication have received European Union (EU) and United States (US), and/or Japan (JP) marketing approval on or after 01 January 2014 or by the US or EU or JP Health Authorities when regulatory submissions in all regions are not planned and after the primary study results have been accepted for publication.
Access Criteria: Formal request from qualified scientific and medical researchers on IPD and clinical study documents from clinical trials supporting products submitted and licensed in the United States, the European Union and/or Japan from 01 January 2014 and beyond for the purpose of conducting legitimate research. This must be consistent with the principle of safeguarding study participants' privacy and consistent with provision of informed consent.
URL: https://vivli.org/ourmember/daiichi-sankyo/

REFERENCES:
- [Derived] Levy BP, Felip E, Reck M, Yang JC, Cappuzzo F, Yoneshima Y, Zhou C, Rawat S, Xie J, Basak P, Xu L, Sands J. TROPION-Lung08: phase III study of datopotamab deruxtecan plus pembrolizumab as first-line therapy for advanced NSCLC. Future Oncol. 2023 Jul;19(21):1461-1472. doi: 10.2217/fon-2023-0230. Epub 2023 May 30. PMID 37249038